CLINICAL TRIAL: NCT04511286
Title: Single-Arm Feasibility Study of Exposure-Based Treatment for Undifferentiated Somatic Symptom Disorder
Brief Title: Exposure-Based Treatment for Undifferentiated Somatic Symptom Disorder
Acronym: SOMEX0
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Erland Axelsson, Principal Investigator, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-01740
Record Dates: First submitted 2020-07-18; First posted 2020-08-13 (Actual); Results first posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Somatic Symptom Disorder
Keywords: Exposure; Feasibility

STUDY DESIGN:
Intervention Model Description: Prospective single-group cohort study
Masking Description: Psychological intervention, patient-reported outcomes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Internet-delivered exposure-based treatment (Experimental): Eight weeks of therapist-guided exposure-based treatment delivered via the Internet.
  Interventions: Behavioral: Exposure

INTERVENTIONS:
Behavioral: Exposure — Systematic confrontation with stimuli associated with symptom-related distress, to achieve therapeutic changes in cognitions or behavior

SUMMARY:
This study investigates the feasibility of a general exposure-based treatment protocol that is intended to work for a large variety of patient groups with a clinically significant preoccupation with physical symptoms. This is a prospective single-group study based at Karolinska Institutet, Stockholm, Sweden, where 40 adults with DSM-5 somatic symptom disorder are enrolled in 8 weeks of therapist-guided exposure-based treatment via the Internet. Exposure is based on general principles but tailored to suit the needs of each patient. Outcomes include patient-reported credibility and expectancy, adherence to the treatment protocol, client satisfaction, and negative events. Within-group effects will also be quantified and discussed in relation to the existing literature.

DETAILED DESCRIPTION:
Background:

A substantial portion of patients in routine care suffer from a recurrent preoccupation with physical symptoms, which often leads to substantial suffering and impairment. Exposure-based treatment - where the patient systematically seeks out that which gives rise to unwanted sensations, cognitions, or behavior - has been found to lead to beneficial effects in several types of symptom preoccupation. Yet, this form of treatment is rarely offered in routine care. This may be partially because existing treatment protocols have been developed for specific symptom clusters (e.g., functional somatic syndromes such as irritable bowel syndrome and fibromyalgia) or specific unwanted responses to symptoms (e.g., the fear of having a severe illness), and that many clinics do not have the resources to offer all these specialized protocols in parallel. An alternative approach could be to base exposure treatment on a more general protocol that may be tailored to suit a larger variety of patient groups who suffer from a recurrent preoccupation with physical symptoms. However, it is yet unclear if the use of such a general treatment protocol for symptom preoccupation would be feasible, for example in terms of patient-reported credibility, adherence, identification with the rationale, and general client satisfaction.

Aim:

To investigate the feasibility of delivering exposure-based treatment using a general protocol for clinically significant symptom preoccupation, without selecting patients based on any specific symptom cluster (such as a functional somatic syndrome) or specific unwanted response to physical symptoms (such as a frequent fear of illness).

Design:

This is a prospective single-group feasibility study based at Karolinska Institutet, Stockholm, Sweden, where 40 adults with somatic symptom disorder according to the Diagnostic and statistical manual of mental disorders 5 (DSM-5) are enrolled in 8 weeks of therapist-guided exposure-based treatment that is delivered via the Internet. Various aspects of feasibility are assessed; most notably: patient-reported credibility and expectancy, adherence to the treatment protocol, client satisfaction, and negative events. Within-group effects are also quantified.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 somatic symptom disorder
* Interest in 8-week intensive psychological treatment to reduce distress and the impact of physical symptoms
* At least 18 years old
* Living in Sweden
* Fluent in Swedish
* Complete pre-treatment assessment

Exclusion Criteria:

* Preoccupation with physical symptoms better explained by another psychiatric condition such as illness anxiety disorder, panic disorder, or obsessive-compulsive disorder
* Severe psychiatric condition, such as bipolar disorder, suicidal ideation, or psychosis
* Medical risks associated with participating in exposure-based treatment, or somatic condition - or treatment for somatic condition - that is an obstacle to participating in exposure-based treatment
* Non-stable continuous pharmacotherapy (dosage changed during the past 4 weeks) and the drug is likely to affect outcome measures (primarily: antidepressants, anticonvulsants, benzodiazepines, nonbenzodiazepines, opioids)
* Alcohol or substance use that is a clear obstacle to therapy
* Planned absence for more than 1 week of the treatment period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erland Axelsson, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
We are willing to consider reasonable requests for individual participant data (IPD) and to consult the responsible parties accordingly. However, we do not expect to be granted permission to share IPD as long as, under Swedish and European Union (EU) data protection and privacy legislation, the IPD constitutes personal data meaning that it is possible to, using the study database, link the IPD to an identifiable living natural person.

REFERENCES:
- [Derived] Hybelius J, Gustavsson A, Af Winklerfelt Hammarberg S, Toth-Pal E, Johansson R, Ljotsson B, Axelsson E. A unified Internet-delivered exposure treatment for undifferentiated somatic symptom disorder: single-group prospective feasibility trial. Pilot Feasibility Stud. 2022 Jul 19;8(1):149. doi: 10.1186/s40814-022-01105-0. PMID 35854392

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We originally aimed to recruit 40 participants for 80% power in two-sided tests of moderate effects (d=0.5) on efficacy outcomes measured at two time points, given a 5% alpha and 15% missing data at post-treatment. In light of the high data retention, prior to the data analysis, we ended the recruitment with 33 participants included in November 2020.
Pre-assignment Details: All participants were enrolled in treatment.
Period: Overall Study
Arm/Group | Internet-delivered Exposure-based Treatment
Started | 33 (First enrollment 2020/11/09)
Completed | 32 (Completed the post-treatment and follow-up assessments, last on 2021/24/02)
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Internet-delivered Exposure-based Treatment
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 33
University education [Count of Participants; unit: Participants] | 27
Employment [Count of Participants; unit: Participants]
  Working full-time | 21
  Working part-time (<90%) | 7
  Retired | 4
  Student | 1

OUTCOME MEASURES:

1. Primary Outcome: Feasibility 1: Distribution of Physical Symptoms
Description: According to the Patient Health Questionnaire-15 (PHQ-15, theoretical range: 0-30, higher score indicates more distressing physical symptoms)
Time Frame: Pre-treatment assessment (within 2 weeks before treatment)
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Internet-delivered Exposure-based Treatment
Number analyzed (Participants) | 33
score on a scale | 11.8 [3 to 20]

2. Primary Outcome: Feasibility 2: Credibility/Expectancy Based on the Credibility/Expectancy Scale
Description: Theoretical range: 0-50, higher score indicates higher credibility/expectancy
Time Frame: Week 3 of treatment
Population: All participants completed the week 3 assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Internet-delivered Exposure-based Treatment
Number analyzed (Participants) | 33
score on a scale | 34.5 (7.0)

3. Primary Outcome: Feasibility 3: Adherence to the Protocol #1: Percentage Completed Modules in the Sample as a Whole
Description: Preregistered target: at least 60% completed modules in the sample as a whole. In this study, all participants were enrolled in the same type of treatment and were thus offered to work with the same treatment modules. This outcome was the proportion of modules completed in total by all participants, out of the total modules available to all participants.
Time Frame: Adherence data collected over the entire course of the treatment, up to 8 weeks.
Population: In this study, all 33 participants were enrolled in the same type of treatment and were thus offered to work with the same five treatment modules.
Measure: Count of Units; unit: Modules
Units Other Than Participants: Modules
Arm/Group | Internet-delivered Exposure-based Treatment
Number analyzed (Participants) | 33
Number analyzed (Modules) | 165
Modules | 150

4. Primary Outcome: Feasibility 4: Patient-reported Adequacy of Rationale as Assessed Using a Questionnaire Developed Specifically for This Purpose (Theoretical Range: 0-10)
Description: From 0 ("not at all relevant") to 10 ("extremely relevant"). Was originally intended to be administered at week 3, but was administered post-treatment due to an administrative error
Time Frame: Post-treatment assessment (immediately after treatment, completed within 45 days)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Internet-delivered Exposure-based Treatment
Number analyzed (Participants) | 33
score on a scale | 8.4 (1.5)

5. Primary Outcome: Feasibility 5: Adequacy of the Measurement Strategy
Description: Preregistered target: less than 30% missing data at post-treatment, and at least 75% finding the measurement strategy acceptable (less than 7 on a scale from 0 ["Not at all stressful/bothering"] to 10 ["Extremely stressful/bothering"])
Time Frame: Post-treatment assessment (immediately after treatment, completed within 45 days)
Population: Because the question about the measurement strategy was administered at the post-treatment assessment, which was completed by 32/33 participants, 32 was the denominator for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Internet-delivered Exposure-based Treatment
Number analyzed (Participants) | 33
Participants
  Missing data at post-treatment | 1
  Found the measurement strategy acceptable (no cause for distress): number analyzed (Participants) | 32
  Found the measurement strategy acceptable (no cause for distress) | 27

6. Primary Outcome: Feasibility 6: Satisfaction With Treatment as Indicated by a Mean Client Satisfaction Questionnaire (CSQ-8) Score of at Least 22
Description: Theoretical range: 8-32, higher score indicates higher satisfaction. This sum score is based on 8 items, each scored 1-4.
Time Frame: Post-treatment assessment (immediately after treatment, completed within 45 days)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Internet-delivered Exposure-based Treatment
Number analyzed (Participants) | 32
score on a scale | 25.3 (4.7)

7. Primary Outcome: Feasibility 7a: Adverse Events Measured Using Free-text Items #1: Total Number of Reported Events
Description: The respondent was instructed to describe up to three adverse events.
Time Frame: Post-treatment assessment (immediately after treatment, completed within 45 days)
Measure: Number; unit: adverse events
Arm/Group | Internet-delivered Exposure-based Treatment
Number analyzed (Participants) | 32
adverse events | 6

8. Primary Outcome: Feasibility 7b: Adverse Events Measured Using the 20-item Negative Effects Questionnaire (NEQ-20)
Description: Theoretical range: 0-80, higher score indicates more severe adverse events
Time Frame: Post-treatment assessment (immediately after treatment, completed within 45 days)
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Internet-delivered Exposure-based Treatment
Number analyzed (Participants) | 32
score on scale | 5.7 (8.2)

9. Primary Outcome: Feasibility 3: Adherence to the Protocol #2: Percentage of Participants Completing at Least 2 Exposure Exercises
Description: Preregistered target: at least 50% of participants completing at least 2 exposure exercises
Time Frame: Adherence data collected over the entire course of the treatment, up to 8 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Internet-delivered Exposure-based Treatment
Number analyzed (Participants) | 33
Participants | 32

10. Primary Outcome: Feasibility 7a: Adverse Events Measured Using Free-text Items #2: Number of Participants Who Reported at Least One Adverse Event
Description: The respondent was instructed to describe up to three adverse events.
Time Frame: Post-treatment assessment (immediately after treatment, completed within 45 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Internet-delivered Exposure-based Treatment
Number analyzed (Participants) | 32
Participants | 5

11. Secondary Outcome: Patient Health Questionnaire-15 (PHQ-15)
Description: Change pre-post, as derived from linear mixed effects regression models fitted by maximum likelihood estimation using data from all 33 participants, and fitted on all 11 measurement points over the treatment phase (from pre-treatment to post-treatment). Theoretical range: 0-30, higher score indicates more distressing physical symptoms
Time Frame: Screening, pre-treatment assessment (within 2 weeks before treatment), weekly during treatment, Post-treatment assessment (immediately after treatment, completed within 45 days), 3 months after treatment
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Internet-delivered Exposure-based Treatment
Number analyzed (Participants) | 33
units on a scale | -4.2 [-5.5 to -2.9]

12. Secondary Outcome: Somatic Symptom Disorder-B Criteria Scale (SSD-12)
Description: Change pre-post, as derived from linear mixed effects regression models fitted by maximum likelihood estimation using data from all 33 participants, and fitted on all 11 measurement points over the treatment phase (from pre-treatment to post-treatment). Theoretical range: 0-48, higher score indicates higher degree of preoccupation with symptoms
Time Frame: as for outcome 11
Measure: Mean (95% Confidence Interval); unit: Likert scale units
Arm/Group | Internet-delivered Exposure-based Treatment
Number analyzed (Participants) | 33
Likert scale units | -13.0 [-16.5 to -9.4]

13. Secondary Outcome: Symptom Preoccupation Scale (Preliminary Scale)
Description: Under development, higher score indicates higher degree of preoccupation with symptoms. This is to be regarded as an item pool that will be further analyzed in 2024-2025, and in conjunction with data from other clinical trials. As of September 2023, it is therefore not yet possible to provide a theoretical range for this scale, and it is also not possible to provide outcomes.
Time Frame: as for outcome 11
Reporting Status: Not Posted, anticipated posting 2025-06

14. Secondary Outcome: 14-item Health Anxiety Inventory (HAI-14)
Description: Change pre-post, as derived from linear mixed effects regression models fitted by maximum likelihood estimation using data from all 33 participants, and fitted on all 11 measurement points over the treatment phase (from pre-treatment to post-treatment). Theoretical range: 0-42, higher score indicates more health anxiety
Time Frame: Screening, pre-treatment assessment (within 2 weeks before treatment), Post-treatment assessment (immediately after treatment, completed within 45 days), 3 months after treatment
Measure: Mean (95% Confidence Interval); unit: Likert scale units
Arm/Group | Internet-delivered Exposure-based Treatment
Number analyzed (Participants) | 33
Likert scale units | -6.7 [-9.3 to -4.2]

15. Secondary Outcome: Anxiety Sensitivity Index (ASI)
Description: Change pre-post, as derived from linear mixed effects regression models fitted by maximum likelihood estimation using data from all 33 participants, and fitted on all 11 measurement points over the treatment phase (from pre-treatment to post-treatment). Theoretical range: 0-64, higher score indicates more anxiety sensitivity
Time Frame: Screening, pre-treatment assessment (within 2 weeks before treatment), post-treatment assessment Post-treatment assessment (immediately after treatment, completed within 45 days), 3 months after treatment
Measure: Mean (95% Confidence Interval); unit: Likert scale units
Arm/Group | Internet-delivered Exposure-based Treatment
Number analyzed (Participants) | 33
Likert scale units | -9.5 [-13.1 to -6.0]

16. Secondary Outcome: GAD-7
Description: Change pre-post, as derived from linear mixed effects regression models fitted by maximum likelihood estimation using data from all 33 participants, and fitted on all 11 measurement points over the treatment phase (from pre-treatment to post-treatment). Theoretical range: 0-21, higher score indicates more general anxiety
Time Frame: Pre-treatment assessment (within 2 weeks before treatment), post-treatment assessment Post-treatment assessment (immediately after treatment, completed within 45 days), 3 months after treatment
Measure: Mean (95% Confidence Interval); unit: Likert scale units
Arm/Group | Internet-delivered Exposure-based Treatment
Number analyzed (Participants) | 33
Likert scale units | -3.4 [-5.0 to -1.7]

17. Secondary Outcome: Patient Health Questionnaire (PHQ-9)
Description: Change pre-post, as derived from linear mixed effects regression models fitted by maximum likelihood estimation using data from all 33 participants, and fitted on all 11 measurement points over the treatment phase (from pre-treatment to post-treatment). Theoretical range: 0-27, higher score indicates more symptoms of depression
Time Frame: Screening, pre-treatment assessment (within 2 weeks before treatment), weekly during treatments (suicidality), post-treatment assesment (immediately after treatment, completed within 45 days), 3 months after treatment
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Internet-delivered Exposure-based Treatment
Number analyzed (Participants) | 33
units on a scale | -3.2 [-4.6 to -1.8]

18. Secondary Outcome: 12-item WHO Disability Assessment Schedule 2.0 (WHODAS 2.0)
Description: Change pre-post, as derived from linear mixed effects regression models fitted by maximum likelihood estimation using data from all 33 participants, and fitted on all 11 measurement points over the treatment phase (from pre-treatment to post-treatment). Theoretical range: 0-100, higher score indicates more disability
Time Frame: as for outcome 14
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Internet-delivered Exposure-based Treatment
Number analyzed (Participants) | 33
units on a scale | -8.8 [-13.0 to -4.6]

19. Secondary Outcome: Alcohol Use Disorders Identification Test (AUDIT)
Description: Theoretical range: 0-40, higher score indicates more problematic alcohol use
Time Frame: Screening only
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Internet-delivered Exposure-based Treatment
Number analyzed (Participants) | 33
score on a scale | 4.7 (5.7)

20. Secondary Outcome: Drug Use Disorders Identification Test (DUDIT)
Description: Theoretical range: 0-44, higher score indicates more problematic substance use
Time Frame: Screening only
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Internet-delivered Exposure-based Treatment
Number analyzed (Participants) | 33
score on a scale | 0.2 (0.8)

21. Secondary Outcome: Working Alliance Inventory (WAI)
Description: Theoretical range: 6-42, higher score indicates better relationship with the therapist
Time Frame: Week 3 of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Internet-delivered Exposure-based Treatment
Number analyzed (Participants) | 33
score on a scale | 35.2 (5.7)

ADVERSE EVENTS:
Time Frame: 8-week treatment period
Description: We assessed adverse events using free-text items where the respondent was instructed to describe up to three adverse events and rate how much this affected them at the time it occurred and at post treatment. We also administered the 20-item Negative Efects Questionnaire (NEQ-20).
  The reason why 32 (not 33) is reported as the number at risk for the "other" subtype of adverse events is that these data were derived from a post-treamtent questionnaire that was completed by 32/33 participants.
Arm/Group | Internet-delivered Exposure-based Treatment
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 5/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Internet-delivered Exposure-based Treatment (N=32)
increased anxiety, stress or distress (Psychiatric disorders) | 3 — self-reported, free text item
a negative outlook on the future caused by poor treatment outcome (Psychiatric disorders) | 1 — self-reported, free text item
distress caused by conflicting information on how to optimise the effect of meditation (Psychiatric disorders) | 1 — self-reported, free text item

LIMITATIONS AND CAVEATS:
The lack of a control group implies that we cannot determine if change in the efficacy outcomes were caused by participants engaging in exposure. Within-group effects were probably on the conservative side, considering the covid-19 restrictions. Another limitation is that, for pragmatic reasons, the participants were self-selected, which could indicate a highly motivated sample. Moreover, the participants were highly educated with a low average level of functional impairment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/86/NCT04511286/Prot_SAP_000.pdf